CLINICAL TRIAL: NCT02298881
Title: Diversity and Dynamic Stability of the Ocular Surface Microbiome
Brief Title: Ocular Surface Microbiome
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Russell Van Gelder, Professor of Ophthalmology, University of Washington
Other Study IDs: 43018; 1R01EY022038-01A1 (NIH)
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye; Microbiome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swab or scrapings of the cornea
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dry eye group: People with dry eye symptoms
- Non-dry eye group: People with no dry eye symptoms

SUMMARY:
The purpose of this study is to collect samples from the surface of eyelids to try to grow and identify bacteria or fungus that might be present, and to try to understand why people have dry eye symptoms.

DETAILED DESCRIPTION:
"Dry eye" is a very common eye condition, which may or may not be caused by specific microorganisms that live on the surface of the eye. In this study, a combination of tissue culture and molecular biology techniques will be used to identify every microbe (bacteria, fungus, or virus) on the surface of eyes of people with dry eye syndrome, as well as a 'control' group of people who don't have dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ocular surface discomfort with an Ocular Surface Disease Index score of greater than 60
* Subjects with and Ocular Surface disease Index score less than 30
* Males and females age 18 or older

Exclusion Criteria:

* Contact lens wear
* Use of oral or topical antibiotics in past 6 months
* Use of prescription eye medication in past 6 months
* Penetrating ocular or keratoplasty surgery in last 12 months
* Children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients from the investigators' practices at the University of Washington Eye Institute
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
To catalog the bacteria and other micro-organisms that are naturally found on the eye surface. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell N VanGelder, MD, PhD, Principal Investigator — UW Medicine Eye Institute
Locations (1):
- UW Medicine Eye Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Doan T, Akileswaran L, Andersen D, Johnson B, Ko N, Shrestha A, Shestopalov V, Lee CS, Lee AY, Van Gelder RN. Paucibacterial Microbiome and Resident DNA Virome of the Healthy Conjunctiva. Invest Ophthalmol Vis Sci. 2016 Oct 1;57(13):5116-5126. doi: 10.1167/iovs.16-19803. PMID 27699405